CLINICAL TRIAL: NCT03724526
Title: Text Messaging and Cardiovascular Health in Diabetes Mellitus: A Randomized, Controlled Clinical Trial (TEACH Study)
Brief Title: Text Messaging and Cardiovascular Health in Diabetes Mellitus
Acronym: TEACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Huijie Zhang, Clinical Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NFEC-2018-117
Record Dates: First submitted 2018-10-23; First posted 2018-10-30 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus; cardiovascular disease; text message
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: The eligible participants will be randomly allocated into intervention and control groups in a 1:1 ratio. The intervention group will receive text messages in addition to usual care for 12 months, while the control group will receive usual care.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The study is a two-arm, parallel, randomized clinical trial. The primary outcome and secondary outcomes was measured by blinded assessors throughout the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention-Text messaging (Experimental): Participates will receive regular 6 text messages per week for 12 months. They will receive one general education about diabetes and CVD messages, one glucose control message, one blood pressure control message, one healthy eating message, one medication adherence message and one physical activity message per week. Each message will be sent on 6 of 7 randomly selected weekdays and arrived at random times the day during working hours.
  Interventions: Behavioral: Text messaging
- Control (No Intervention): Participates in control group will not receive text messages.

INTERVENTIONS:
Behavioral: Text messaging — Intervention-Text messaging: Participants will receive regular text messages for 12 months. Each participant will receive 6 text messages per week. They will receive one general education about diabetes and CVD messages, one glucose control message, one blood pressure control message, one healthy eating message, one medication adherence message and one physical activity message per week.
  Control: The control group will receive the usual care.
  Arms: Intervention-Text messaging

SUMMARY:
The purpose of the study of the proposed randomized trial is to evaluate the effectiveness of automated mobile phone text message-based intervention in improving lifestyle modification, medication adherence and CVD risk factors (glycated hemoglobin [HbA1C], systolic blood pressure [SBP], and LDL-cholesterol) over 12 months among patients with type 2 diabetes.

DETAILED DESCRIPTION:
Most patients with diabetes have multiple risk factors, such as obesity, hypertension, and dyslipidemia, or with arteriosclerotic cardiovascular disease (ASCVD). The purpose of the study of the proposed randomized trial will examine the effect of health text messages in improving lifestyle modification, medication adherence and CVD risk factors (glycated hemoglobin [HbA1C], systolic blood pressure [SBP], and LDL-cholesterol) over 12 months among patients with type 2 diabetes. This study is a multicenter prospective, randomized, controlled clinical trial. The eligible participants will be randomly allocated into intervention and control groups in a 1:1 ratio. The intervention group will receive text messages in addition to usual care for 12 months, while the control group will receive usual care. The messages will target lifestyle recommendation, glucose control, blood pressure control, healthy eating, medication adherence, physical activity and smoking cessation. Each message will be sent on 6 of 7 randomly selected weekdays and arrived at random times the day during working hours. The primary outcome is the combined changes in HbA1C, SBP and LDL-cholesterol levels, simultaneous modeled using a scaled marginal model. The Secondary outcome includes the net change of CVD risk factors (glycated hemoglobin [HbA1C], systolic blood pressure [SBP], and LDL-cholesterol), and the proportion of participants with HbA1C <7% (<7.5% if with clinical CVD), BP<140/90 mm Hg, and LDL-cholesterol <100 mg/dL, and net change in estimated 10-year risk of CHD and CVD. The primary outcome and secondary outcome will be measured at month 3, 6, and 12 visits.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18 years and over
2. Patients with poorly controlled type 2 diabetes who are undergoing routine treatment (defined as HbA1c≥ 7% or HbA1c≥7.5% if combined with clinical cardiovascular disease) have at least one risk factor for other cardiovascular disease (SBP≥140 mmHg and/or DBP≥90 mmHg and/or low density lipoprotein cholesterol≥100mg/dL) or clinical atherosclerotic cardiovascular disease (acute coronary syndrome, ischemic stroke transient ischemic attack or peripheral arterial disease)
3. Participants can provide written informed consent.
4. Participants required access to a smartphone, and be able to receive and read text message.

Exclusion Criteria:

1. Participants were in functional New York Heart Association class III or IV, and were on haemodialysis;
2. Pregnant women or women planning to become pregnant
3. Participants cannot be followed up for 12 months (due to health status or migration)
4. Participants cannot provide written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 819 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Combined changes in HbA1C, SBP and LDL-cholesterol levels, simultaneous modeled using a scaled marginal model. | 12 months

SECONDARY OUTCOMES:
Change in glucose level measured by HbA1C level | 12 months
Change in Systolic blood pressure level | 12 months
Change in LDL-cholesterol level | 12 months
The proportion achieving levels of Hba1c < 7% (< 7.5% if combined with cardiovascular disease) | 12 months
The proportion achieving levels of blood pressure <140/90 mm Hg | 12 months
The proportion achieving levels of LDL-cholesterol <100 mg/dL | 12 months
Change in Framingham Risk Score | 12 months
Change in ACC/AHA Risk Score of CVD | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Huijie Zhang, M.D.&Ph.D, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang PZ, Guo D, Liu CQ, Chen N, Liu JF, Lei XZ, Yang LJ, Liu YT, Li X, Huang JF, Du CM, Wang K, Mo W, Lin JY, Huang CS, Xu BY, Wei XY, Liu DY, Huang JL, Huang Y, Xue YM, Zeng YM, Liu SQ, Ma ZM, Zhang HJ. Mobile App-Based Intervention and Cardiovascular Risk Factors in Patients With Uncontrolled Type 2 Diabetes: A Randomized Clinical Trial. JAMA Netw Open. 2025 Sep 2;8(9):e2529762. doi: 10.1001/jamanetworkopen.2025.29762. PMID 40892411